CLINICAL TRIAL: NCT02321514
Title: Expanded Clinical Study of the Tendyne Mitral Valve System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-03
Record Dates: First submitted 2014-12-10; First posted 2014-12-22 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Mitral Valve Regurgitation
Keywords: ABT-CIP-10337; Tendyne Bioprosthetic Mitral Valve System
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Tendyne Mitral Valve System (Experimental): Patients will undergo transcatheter mitral valve replacement
  Interventions: Device: Tendyne Mitral Valve System

INTERVENTIONS:
Device: Tendyne Mitral Valve System — Patients will undergo transcatheter mitral valve replacement using Tendyne Mitral Valve system

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Tendyne Mitral Valve System in the treatment of severe mitral regurgitation in patents with functional disability greater than or equal to NYHA Class II, who are not suitable candidates for surgical replacement with otherwise available devices. Follow-up evaluations will be conducted through 5 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Severe mitral regurgitation of primary or secondary etiology according to MVARC (Mitral Valve Academic Research Consortium) 2015 defined as:

   * For Degenerative MR: EROA ≥ 40 mm^2 or regurgitant volume ≥ 60ml
   * For Secondary MR: EROA ≥ 20 mm^2 or regurgitant volume ≥ 30ml
2. New York Heart Association (NYHA) functional Class ≥ II while on guideline directed medical therapy (GMDT), including device therapy (CRT) if indicated.
3. Heart team determines patient is not a suitable candidate for traditional surgical treatment according to valid guidelines.
4. Age 18 years or older.

Exclusion Criteria:

1. Severe mitral annular calcification, severe mitral stenosis, valvular vegetation or mass.
2. Left Ventricle (LV) or Left Atrium (LA) thrombus.
3. Patient has a chest condition that prevents transapical access.
4. Left ventricular ejection fraction (LVEF) less than 30% by echocardiogram.
5. Left Ventricular End Diastolic Diameter (LVEDD) > 7.0 cm.
6. Prior surgical or interventional treatment of mitral or aortic valves (e.g. valve repair or replacement, MitraClip, edge to edge repair, aortic balloon valvuloplasty, etc.).
7. Any planned surgery or interventional procedure within the period of 30 days prior to 30 days following the implant procedure. This includes any planned concomitant cardiovascular procedure such as PCI, pulmonary vein ablation, left atrial appendage occlusion, septal defect repair, etc.
8. Cardiac resynchronization therapy device or implantable pulse generator implanted within three months of planned implant procedure.
9. Myocardial Infarction (MI) within 30 days of the planned implant procedure.
10. Symptomatic, unresolved multi-vessel coronary artery disease (CAD) or unprotected left main coronary artery disease requiring stenting or Coronary Artery Bypass Grafting (CABG).
11. Cerebrovascular accident (CVA) within six months of planned implant procedure.
12. Unresolved severe symptomatic carotid stenosis (> 70% by ultrasound).
13. Cardiogenic shock or hemodynamic instability requiring inotropes or mechanical support devices at the time of planned implant procedure.
14. Severe tricuspid regurgitation, tricuspid valve disease requiring surgery or severe right ventricular dysfunction.
15. Hypertrophic or restrictive cardiomyopathy, constrictive pericarditis or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology.
16. Any of the following: leukopenia, acute anemia, thrombocytopenia, history of bleeding diathesis, or coagulopathy if cannot be adequately treated.
17. History of endocarditis within six months of planned implant procedure.
18. Active systemic infection requiring antibiotic therapy.
19. Known hypersensitivity or contraindication to procedural or post-procedural medications (e.g., contrast solution, anti-coagulation therapy) which cannot be adequately managed medically or hypersensitivity to nickel or titanium.
20. Patient is undergoing hemodialysis due to chronic renal failure.
21. Patient has pulmonary arterial hypertension (fixed PAS >70mmHg).
22. Patient has COPD and is on home oxygen.
23. Patient refuses blood transfusions.
24. Pregnant, lactating, or planning pregnancy within next 12 months.
25. Participating or planning participation in an investigational drug or another device study.
26. Patient or legal guardian unable or unwilling to give informed consent.
27. Patient unable or unwilling to comply with study required testing and follow-up visits.
28. Patients with non-cardiac co-morbidities that are likely to result in a life expectancy of less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2025-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (13):
  - Honor Health Scottsdale Shea Medical Center, Scottsdale, Arizona
  - MedStar Washington Hospital, Washington D.C., District of Columbia
  - Morton Plan Mease Health Care, Clearwater, Florida
  - Delray Medical Center, Delray Beach, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northshore University Health System, Evanston, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - St. Francis Hospital, Roslyn, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pinnacle Health - Harrisburg Hospital, Harrisburg, Pennsylvania
  - Baylor Heart & Vascular Center, Dallas, Texas
  - West Virginia University, Morgantown, West Virginia
- Australia (3):
  - Flinders Medical Center, Bedford Park
  - Prince Charles Hospital, Chermside
  - St. Vincent's Hospital, Sydney
- France (5):
  - Bordeaux University Hospital, Bordeaux
  - CHRU de Lille, Lille
  - Lyon University Hospital, Lyon
  - Rennes University Hospital, Rennes
  - Clinique Pasteur, Toulouse
- Germany (9):
  - Deutsche Herzzentrum Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - University Hospital Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - University Heart Center Hamburg, Hamburg
  - Leipzig Heart Center, Leipzig
  - University Medical Center Mainz, Mainz
  - Ludwig-Maximilians-Universität München (LMU), Munich
  - University of Rostock, Rostock
- Italy (5):
  - Ospedale Ferrarotta - Catania, Catania
  - San Raffaele, Milan
  - Pisa University, Pisa
  - Humanitas Research Hospital, Rozzano
  - San Donato, San Donato Milanese
- St. Antonius Hospital, Nieuwegein, Netherlands
- Oslo University Hospital, Oslo, Norway
- Karolinksa University Hospital, Solna, Sweden
- University Hospital of Zurich, Zurich, Switzerland
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Muller DWM, Sorajja P, Duncan A, Bethea B, Dahle G, Grayburn P, Babaliaros V, Guerrero M, Thourani VH, Bedogni F, Denti P, Dumonteil N, Modine T, Jansz P, Chuang ML, Blanke P, Leipsic J, Badhwar V. 2-Year Outcomes of Transcatheter Mitral Valve Replacement in Patients With Severe Symptomatic Mitral Regurgitation. J Am Coll Cardiol. 2021 Nov 9;78(19):1847-1859. doi: 10.1016/j.jacc.2021.08.060. PMID 34736561
- [Derived] Muller DWM, Farivar RS, Jansz P, Bae R, Walters D, Clarke A, Grayburn PA, Stoler RC, Dahle G, Rein KA, Shaw M, Scalia GM, Guerrero M, Pearson P, Kapadia S, Gillinov M, Pichard A, Corso P, Popma J, Chuang M, Blanke P, Leipsic J, Sorajja P; Tendyne Global Feasibility Trial Investigators. Transcatheter Mitral Valve Replacement for Patients With Symptomatic Mitral Regurgitation: A Global Feasibility Trial. J Am Coll Cardiol. 2017 Jan 31;69(4):381-391. doi: 10.1016/j.jacc.2016.10.068. Epub 2016 Dec 28. PMID 28040318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 191 patients were enrolled and attempted TMVR procedure with Tendyne Mitral Valve System. The first subject was implanted on 24 November 2014. The last subject was implanted on 02 June 2020 and completed the 1-month follow-up evaluation on July 6, 2020.
Groups:
- Tendyne Mitral Valve System: Tendyne Mitral Valve System
  Patients will undergo transcatheter mitral valve replacement using Tendyne Mitral Valve system
Period: Overall Study
Arm/Group | Tendyne Mitral Valve System
Started | 191
Completed | 166
Not Completed | 25
Not completed — Death | 15
Not completed — Missed Visit | 7
Not completed — Study Exit | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tendyne Mitral Valve System
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants were identified in both Race and Ethnicity
  Participants
    Hispanic or Latino | 3
    Not Hispanic or Latino | 185
    Caucasian | 177
    Asian | 5
    Black or African American | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 24
  France | 18
  Germany | 22
  Italy | 20
  Netherlands | 3
  Norway | 10
  Sweden | 1
  Switzerland | 1
  United Kingdom | 18
  United States | 74
NYHA Class, III/IV [Count of Participants; unit: Participants] — NYHA functional classification system relates symptoms to everyday activities and the patient's quality of life.
  NYHA Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  NYHA Class II: Subjects with cardiac disease resulting in slight limitation of physical activity.
  NYHA Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  NYHA Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Participants | 133

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Number of Participants With Composite of Device Success and Freedom From Device or Procedure Related Serious Adverse Events (SAEs)
Description: Device success and freedom from the following device- or procedure-related serious adverse events (SAEs) at 30 days post the index procedure, will be classified by the Clinical Events Committee (CEC):
  * Cardiovascular death
  * Reintervention caused by valve-related dysfunction
  * Disabling stroke
  * Myocardial infarction (MI)
  * Life-threatening bleeding (BARC Type 2, 3, and 5)
  * Major Vascular Complications
  * Renal failure requiring dialysis
  * Other device-related SAEs
  * Other procedure-related SAEs
Time Frame: 30 days post-index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Tendyne Mitral Valve System
Number analyzed (Participants) | 170
Participants | 120

2. Primary Outcome: Performance Endpoint: Number of Participants With MR Grade ≤ 2
Description: Proportion of subjects with mitral regurgitation (MR) grade ≤ 2, per echocardiography core laboratory will be assessed.
  MR severity is graded on a scale of 0+ to 4+ where 0+ means absence of mitral regurgitation, 1+ is mild, 2+ is moderate, 3+ is moderate-to-severe and 4+ is severe.
Time Frame: 30 days post-index procedure
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Tendyne Mitral Valve System
Number analyzed (Participants) | 158
Participants | 158

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Tendyne Mitral Valve System
All-Cause Mortality (participants affected / at risk) | 15/191
Serious Adverse Events (participants affected / at risk) | 117/191
Other Adverse Events (participants affected / at risk) | 123/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tendyne Mitral Valve System (N=191)
Atrial fibrillation (Cardiac disorders) | 9
Bleeding complications (Vascular disorders) | 1
Blood loss requiring transfusion (Vascular disorders) | 12
Cardiac Arrest (Cardiac disorders) | 6
Cardiac Arrhythmia (Cardiac disorders) | 8
Cardiac tamponade (Cardiac disorders) | 1
Conduction defect/cardiac arrhythmia (Cardiac disorders) | 2
Decreased LV function and/or cardiac output (Cardiac disorders) | 5
Device erosion, migration or malposition (Cardiac disorders) | 3
Dizziness (Cardiac disorders) | 1
Endocarditis (Cardiac disorders) | 1
Heart Failure (Cardiac disorders) | 2
Heart Failure, Worsening (Cardiac disorders) | 19
Hypotension (Cardiac disorders) | 9
Infection (Cardiac disorders) | 2
Mitral valve regurgitation, worsening (Cardiac disorders) | 1
Multiple Organ Failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Pain (Cardiac disorders) | 1
Paravalvular leak (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Pleural Effusion (Cardiac disorders) | 4
Pulmonary edema (Cardiac disorders) | 1
Sepsis (Cardiac disorders) | 1
Shock (Cardiac disorders) | 12
Tachycardia (Cardiac disorders) | 1
Thrombosis, Device (Cardiac disorders) | 3
Vascular & access-related complications (Vascular disorders) | 4
Vascular & access-related complications - Transapical (Vascular disorders) | 3
Other - Cardiovascular (Cardiac disorders) | 3
Blood loss not requiring transfusion (Skin and subcutaneous tissue disorders) | 1
Vascular & access-related complications (Skin and subcutaneous tissue disorders) | 1
Abnormal lab values (Metabolism and nutrition disorders) | 1
Renal insufficiency or failure (Metabolism and nutrition disorders) | 1
Blood loss requiring transfusion (Gastrointestinal disorders) | 4
Cardiac Arrest (Gastrointestinal disorders) | 1
Liver failure (Gastrointestinal disorders) | 2
Nausea/Vomiting (Gastrointestinal disorders) | 1
Pain (Gastrointestinal disorders) | 1
Sepsis (Gastrointestinal disorders) | 1
Other - Gastrointestinal/Digestive (Gastrointestinal disorders) | 3
Other - Genitourinary (Gastrointestinal disorders) | 1
Renal insufficiency or failure (Renal and urinary disorders) | 14
Urinary Tract Infection (Renal and urinary disorders) | 3
Other - Genitourinary (Renal and urinary disorders) | 1
Blood loss not requiring transfusion (General disorders) | 1
HEENT- Blood loss not requiring transfusion (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 7
Blood loss not requiring transfusion (Blood and lymphatic system disorders) | 1
Blood loss requiring transfusion (Blood and lymphatic system disorders) | 14
Hemolysis (Blood and lymphatic system disorders) | 1
Infection (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Shock (Blood and lymphatic system disorders) | 1
Supratherapeutic INR (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Other - Cytokine reaction (Blood and lymphatic system disorders) | 1
Other - Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Altered mental status (Nervous system disorders) | 1
Embolism, Other (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 2
Other - Neurologic (Nervous system disorders) | 3
Altered mental status (Psychiatric disorders) | 1
Blood loss requiring transfusion (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac Arrest (Respiratory, thoracic and mediastinal disorders) | 1
Heart Failure, Worsening (Respiratory, thoracic and mediastinal disorders) | 2
Infection (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 14
Respiratory Difficulty (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory Insufficiency/Failure (Respiratory, thoracic and mediastinal disorders) | 11
Sepsis (Respiratory, thoracic and mediastinal disorders) | 1
Other - Respiratory (Respiratory, thoracic and mediastinal disorders) | 5
Altered mental status (General disorders) | 1
Anemia (General disorders) | 1
HEENT- Blood loss requiring transfusion (General disorders) | 1
Fever (General disorders) | 1
Infection (General disorders) | 1
Liver failure (General disorders) | 1
Multiple Organ Failure (General disorders) | 1
Pleural Effusion (General disorders) | 1
Renal insufficiency or failure (General disorders) | 3
Sepsis (General disorders) | 1
Vascular & access-related complications (General disorders) | 1
Other - Coagulopathy- clotting disorder (General disorders) | 1
Other - Increased CT output (General disorders) | 1
Other - thoracic drainage (General disorders) | 1
Other - unable to remove chest tube (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tendyne Mitral Valve System (N=191)
Atrial fibrillation (Cardiac disorders) | 16
Cardiac Arrhythmia (Cardiac disorders) | 16
Decreased LV function and/or cardiac output (Cardiac disorders) | 11
Hypotension (Cardiac disorders) | 19
Paravalvular leak (Cardiac disorders) | 14
Abnormal lab values (Metabolism and nutrition disorders) | 10
Fever (Metabolism and nutrition disorders) | 14
Other - Gastrointestinal/Digestive (Gastrointestinal disorders) | 11
Renal insufficiency or failure (Renal and urinary disorders) | 16
Anemia (Blood and lymphatic system disorders) | 13
Leukocytosis (Blood and lymphatic system disorders) | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Pain (Musculoskeletal and connective tissue disorders) | 19
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 18
Respiratory Difficulty (Respiratory, thoracic and mediastinal disorders) | 10
Other - Respiratory (Respiratory, thoracic and mediastinal disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02321514/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT02321514/SAP_001.pdf